CLINICAL TRIAL: NCT03904953
Title: Effects of Pilates Training on Respiratory Muscle Strenght in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Pilates; Respiratory muscle strenght
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Clinical pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: Pilates Training
- Control group (Active Comparator): Stretching of erector spine, hip flexors, hamstring muscles and gastro-soleus muscles; back-strengthening of cervical, thoracic and lumbar spine and posture exercises will be taught to the patients in the first session and the patients will be requested to repeat the exercises three times a week for 8 weeks individually at home.
  Interventions: Other: Conventional exercise programme

INTERVENTIONS:
Other: Pilates Training — Clinical pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Arms: Study group
Other: Conventional exercise programme — Stretching of erector spine, hip flexors, hamstring muscles and gastro-soleus muscles; back-strengthening of cervical, thoracic and lumbar spine and posture exercises will be taught to the patients in the first session and the patients will be requested to repeat the exercises three times a week for 8 weeks individually at home.
  Arms: Control group

SUMMARY:
Background: Ankylosing Spondylitis (AS) is a chronic, inflammatory rheumatic disease that effects primarily axial-spine. Reduction of flexibility and mobility is important factors that can cause muscle weakness, impairment quality of life, reduction of exercise tolerance and pulmonary capacity with the progression of AS. The purpose of this study is to investigate the effects of pilates exercises on mobility, quality of life and respiratory muscle strength in patients with AS.

Methods: Forty patients will be included who are aged between 18-55 years and got diagnosed according to Modified New York criterias.Patients will be divided into two groups randomly. Pilates training will be performed to the treatment group and conventional exercises will be performed to the control group during 8 weeks. Respiratory muscle strength, quality of life, spinal mobility, thorax expansion, respiratory functions, physical activity level, exercise capasity and disease activity will be evaluated at first session and at the end of the 8th week in this study.

DETAILED DESCRIPTION:
Objective: Ankylosing Spondylitis (AS) is a chronic, inflammatory rheumatic disease that effects primarily axial-spine. With progression of disease, flexibility of thorax and spine will be get lost. It is reported that mobility, function, respiratory muscle strength and endurance get worse in AS patients. Reduction of flexibility and mobility is important factors that can cause muscle weakness, impairment quality of life, reduction of exercise tolerance and pulmonary capacity with the progression of AS. To writer's knowledge, there has been no study examining the effects of pilates exercises on mobility, function and respiratory muscle strength in AS patients. The purpose of this study is to investigate the effects of pilates exercises on mobility, function and respiratory muscle strength in patients with AS.

Methods: Forty patients were included who are aged between 18-65 years and got diagnosed according to Modified New York criterias. Patients who have incooperation, malignancy and pregnancy will be excluded from the study. Patients will be divided into two groups randomly. Pilates training will be performed to the treatment group and conventional exercises will be performed to the control group during 8 weeks Respiratory muscle strength will be assessed by maximal inspiratory and expiratory pressures. Thorax expansion will be measured from regions of axillar, subcostal and epigastric by tape measure. To evaluate disease activity and spinal mobility, we will use Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Bath Ankylosing Spondylitis Metrology Index (BASMI), respectively. Quality of life will be evaluated with Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL). Exercise capacity will be assessed by 6 minutes walk test. Pilates exercises will be performed 3 days in a week for 8 weeks. Conventional exercise programme will be taugt to the control group and requested to perform them at home. The assessments will be repeated in before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged between 18-55 years,
* Patients who got diagnosed according to Modified New York criteria
* Patients who are being followed at Gazi University Department of Rheumatology.

Exclusion Criteria:

* Patients who have exercise habits
* Incooperation
* Malignancy
* Pregnancy
* Patients who have changes of medical treatment in the last 3 months
* Patients who have another disease that can effect pulmonary functions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-06-02 (Estimated); Study Completion 2019-10-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | 5 minutes
  Respiratory muscle strength will be assessed by digital mouth-pressure meter (Micro Medical MicroRM, Rochester, England). Maksimal inspiratory pressure (MIP) and Maksimal Expiratory Pressure (MEP) will be measured with the subject sitting and breathing through a mouthpiece by encouraged verbally, after clamping the nose (cmH2O). To measure MIP, the patient will be requested to breath in quickly and deeply until total lung capacity, just after breath out maximally until residual volume. To measure MEP, the patient will be requested to breath until total lung capacity and then breath out quickly until residual volume. Leaks around the mouthpiece will be avoided. The best of five attempts will be selected and stated as percent of expected values according to sex and age

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index | 5 minutes
  Spinal mobility will assessed and scored by Bath Ankylosing Spondylitis Metrology Index (BASMI). There are five measurements including lateral lumbar flexion, tragus-to-wall distance, lumbar flexion (Modified Schober), maximal intermalleolar distance and cervical rotation according to the index. Each subscale is scored between 0 and 10. All points are then averaged to calculate total score. Higher values represent worse outcomes.
Ankylosing Spondylitis Quality of Life Questionnaire | 1 minute
  Quality of life will be assessed with Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) which has 18 items, each with response True/Not True. 'True responses are summed to create a total score. High scores mean poor quality of life
Thorax pain | 1 minute
  Visual Analog Scale (VAS) will be used to determine the intensity of thorax pain; 0 means 'no pain' while 10 means 'unbearable pain'.
Chest expansion | 2 minutes
  Chest expansion will be measured with a tape placed circumferentially around the chest wall (axillar, subcostal, epigastric) in cm.
Aerobic capacity | 10 minutes
  Aerobic capacity will be assessed with 6 minute walk test (6MWT) which is a submaximal effort test. 6MWT is a distance required to fast-paced walk on flat floor in length 30 meters. The aim of the 6MWT is to walk as long as the patient can walk in 6 minutes. Dyspnoea and fatigue level are recorded at the end of the test. Distance covered by the patient is calculated at the of 6 minutes
Bath Ankylosing Spondylitis Disease Activity Index | 1 minute
  Bath Ankylosing Spondylitis Disease Activity Index which consists of 6 questions will be used to evaluate disease activity. BASDAI is a composite index, consisting of an assessment on a 10 cm horizontal visual analog scale of fatigue, axial pain, peripheral pain, enthesopathy and stiffness. Fifth and sixth questions are averaged. Addition to this score, other questions are averaged. Total score is between 0 and 10. Higher score represent worse outcome.
International Physical Activity Questionnaire- Short Form | 1 minute
  This questionnaire obtains information about how much time is spent while walking and in moderate and vigorous activities and sitting duration in the last 7 days. The questionnaire records the activity of four intensity levels: 1) vigorous-intensity activity, 2) moderate-intensity activity, 3) walking, and 4) sitting. Durations are multiplied by known METs per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. A sitting question is not included in physical activity score. The questionnaire is scored as: those who score high on the IPAQ engage in vigorous intensity activity of at least 1500 MET minutes a week, those who score modarete on the IPAQ of at least 600 MET minutes a week, those who score a low level of physical activity on the IPAQ means that not meeting any of the criteria for either moderate or high levels of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Study Director — Gazi University Faculty of Health Sciences
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altan L, Korkmaz N, Dizdar M, Yurtkuran M. Effect of Pilates training on people with ankylosing spondylitis. Rheumatol Int. 2012 Jul;32(7):2093-9. doi: 10.1007/s00296-011-1932-9. Epub 2011 Apr 17. PMID 21499876
- [Background] Rosu MO, Topa I, Chirieac R, Ancuta C. Effects of Pilates, McKenzie and Heckscher training on disease activity, spinal motility and pulmonary function in patients with ankylosing spondylitis: a randomized controlled trial. Rheumatol Int. 2014 Mar;34(3):367-72. doi: 10.1007/s00296-013-2869-y. Epub 2013 Sep 26. PMID 24071935